CLINICAL TRIAL: NCT02549430
Title: Phase 2,Open-label,Multicenter,Randomized Study of PD0332991 (Oral CDK4/6 Inhibitor) Monotherapy and in Combination With the HT to Which the pt Has Progressed in the Previous Line for ER+,Her2- Post-menopausal Advanced Breast Cancer Pts
Brief Title: To Reverse ENDocrine Resistance Trial - PD 0332991 Monotherapy vs PD 0332991 in Combination With the Endocrine Therapy
Acronym: TREnd
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Sandro Pitigliani (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TREnd; 2011-005637-38 (EudraCT Number)
Record Dates: First submitted 2015-08-27; First posted 2015-09-15 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: Advanced breast cancer; Postmenopausal; ER positive; Her2 negative
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Anastrozole; Letrozole; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Palbociclib monoterapy
  Interventions: Drug: Palbociclib
- Arm B (Experimental): Palbociclib + HT (Anastrozole, Letrozole, Exemestane, Fulvestrant)
  Interventions: Drug: Palbociclib; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Fulvestrant

INTERVENTIONS:
Drug: Palbociclib — Palbociclib 125 mg/day orally in an ongoing 3:1 schedule (3 weeks on/1 week off)
  Other Names: PD0332991
Drug: Anastrozole — Continuation of prior anastrozole 1mg/day orally in a continuous regimen
  Arms: Arm B
Drug: Letrozole — Continuation of prior letrozole 2.5mg/day orally in a continuous regimen
  Arms: Arm B
Drug: Exemestane — Continuation of prior exemestane 25mg/day orally in a continuous regimen
  Arms: Arm B
Drug: Fulvestrant — Continuation of prior fulvestrant 500mg intramuscular injection every 4 weeks in a continuous regimen
  Arms: Arm B

SUMMARY:
This study aims to assess the activity of PD0332991 in monotherapy and in combination with the endocrine therapy (anastrozole, letrozole, exemestane or fulvestrant) on which the patient has progressed in the previous line for advanced breast cancer in order to reverse endocrine resistance.

DETAILED DESCRIPTION:
In a clinical context, there is a lack of molecular compounds with demonstrated clinical activity in delaying/reversing resistance to endocrine agents. CDK 4/6 inhibitors may represent a biologically-driven option in this context.

With the present study investigators aim to complement the ongoing trial on PD0332991 by acquiring information on its clinical activity in post-menopausal patients with ER positive, Her2 negative advanced breast cancer patients already pretreated with a first-line or second line endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of adenocarcinoma of the breast with evidence of metastatic disease
* ER positive tumor ≥ 10%
* HER2 negative breast cancer by FISH or IHC
* Progression of advanced breast cancer on first or second line endocrine therapy for advanced breast cancer
* Paraffin-embedded tumor available for centralized assessment of biomarkers
* Measurable disease according to RECIST 1.1 (bone only disease is allowed only if measurable).
* Postmenopausal status
* Eastern Cooperative Oncology Group (ECOG) Performance status 0 -2
* Resolution of all acute toxic effects of prior therapy or surgical procedures to CTCAE grade >1
* Adequate organ function

Exclusion Criteria:

* Unstable brain metastases
* Prior treatment with more than one line of CT or more than two lines of HT advanced breast cancer or any CDK inhibitor
* Current treatment with therapeutic doses of anticoagulant
* Current use or anticipated need for food or drugs that are known strong CYP3A4 inhibitors / inducers, drugs that are predominantly metabolized by CYP3A with narrow therapeutic indices, drugs with the potential of prolonging QT interval
* Diagnosis of any secondary malignancy within the last 3 years
* Active inflammatory bowel disease or chronic diarrhea
* Known human immunodeficiency virus infection; active hepatitis C, active hepatitis B

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-10; Primary Completion 2017-02-09 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Incidence of complete response (CR), partial response (PR) or stable disease (SD) ≥24 weeks (clinical benefit) | Baseline up to 3 years
  All randomized patients with adequate baseline disease assessment with measurable disease, the disease under study and who start treatment on the assigned arm will be considered evaluable for clinical benefit (CB). The probability of CB on each randomized treatment arm will be estimated by dividing the number of patients with CB by the number of evaluable patients randomized to the treatment arm.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Baseline up to 3 years
  PFS is the time from randomization date to date of first documentation of progression or death due to any cause, whichever occurs first. Documentation of progression must be by objective disease assessment as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. All patients randomized will be considered evaluable for PFS.
Objective Response (OR) | Baseline up to 3 years
  All randomized patients with adequate baseline disease assessment with measurable disease, the disease under study and who start treatment on the assigned arm will be considered evaluable for objective response (CR or PR). The probability of OR on each randomized treatment arm will be estimated by dividing the number of patients with OR by the number of evaluable patients randomized to the respective treatment arm ("response rate").
Overall Survival (OS) | Baseline up to 6 years
  OS is the time from randomization date to date of death due to any cause. All patients randomized will be considered evaluable for OS.
Time to Progression (TTP) | Baseline up to 3 years
  TTP is the time from randomization date to date of first documentation of objective progression. All patients randomized will be considered evaluable for TTP.
Duration of Response (DR) | Baseline up to 3 years
  For patients with an objective response (CR or PR), duration of response is the time from first documentation of CR or PR to date of first documentation of objective progression or death. Date of first documentation of progression and date of first documentation of CR or PR will be based on investigator assessment of response.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Baseline up to 3 years
  All patients treated with at least one dose of trial treatment will be included in safety analyses. Adverse events will be summarized by treatment and by the frequency of patients experiencing treatment emergent adverse events corresponding to body systems and MedDRA preferred term. Adverse events will be graded by worst NCI CTCAE v4.0 grade.

CONTACTS AND LOCATIONS:
Overall Officials: LUCA MALORNI, MD, Principal Investigator — Azienda USL 4 Prato
Locations (6):
- Italy (6):
  - Azienda Ospedaliera Papa Giovanni Xxiii, Bergamo
  - Ospedale Antonio Perrino, Brindisi
  - Istituto Europeo Oncologia, Milan
  - A.O.U. Federico Ii Di Napoli, Napoli
  - Fondazione Maugeri, Pavia
  - A.O.U. S. Maria Della Misericordia Di Udine, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galardi F, De Luca F, Biagioni C, Migliaccio I, Curigliano G, Minisini AM, Bonechi M, Moretti E, Risi E, McCartney A, Benelli M, Romagnoli D, Cappadona S, Gabellini S, Guarducci C, Conti V, Biganzoli L, Di Leo A, Malorni L. Circulating tumor cells and palbociclib treatment in patients with ER-positive, HER2-negative advanced breast cancer: results from a translational sub-study of the TREnd trial. Breast Cancer Res. 2021 Mar 24;23(1):38. doi: 10.1186/s13058-021-01415-w. PMID 33761970
- [Derived] Malorni L, Curigliano G, Minisini AM, Cinieri S, Tondini CA, D'Hollander K, Arpino G, Bernardo A, Martignetti A, Criscitiello C, Puglisi F, Pestrin M, Sanna G, Moretti E, Risi E, Biagioni C, McCartney A, Boni L, Buyse M, Migliaccio I, Biganzoli L, Di Leo A. Palbociclib as single agent or in combination with the endocrine therapy received before disease progression for estrogen receptor-positive, HER2-negative metastatic breast cancer: TREnd trial. Ann Oncol. 2018 Aug 1;29(8):1748-1754. doi: 10.1093/annonc/mdy214. PMID 29893790